CLINICAL TRIAL: NCT05453487
Title: Immunogenicity and Safety of an Inactivated SARS-CoV-2 Vaccine (Sinopharm BBIBP-CorV) Coadministered With Rabies Vaccine in China: a Multicentre, Randomised, Controlled, Phase 4 Trial
Brief Title: Immunogenicity and Safety of an Inactivated SARS-CoV-2 Vaccine (Sinopharm BBIBP-CorV) Coadministered With Rabies Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Guizhou Center for Disease Control and Prevention (Other); Shaanxi Provincial Center for Disease Control and Prevention (Other); Beijing Institute of Biological Products Co Ltd. (Industry); Changchun Institute of Biological Products Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BBIBP-Cov+Rabies
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Rabies
MeSH Terms: conditions — COVID-19; Rabies | interventions — COVID-19 Vaccines; Rabies Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-Ad group (Experimental): A total of 120 participants received one dose of inactivated COVID-19 vaccine and three doses of rabies vaccine.
  Participants received one dose of inactivated COVID-19 vaccine and rabies vaccine on Day 0, and one dose of rabies vaccine on Day 7 and Day 28.
  Blood sampling was performed on Day 0, Day 28 and Day 42.
  Interventions: Biological: coadministration
- COVID-19 vaccine group (Experimental): A total of 120 participants received one dose of inactivated COVID-19 vaccine on Day 0.
  Blood sampling was performed on Day 0 and Day 28.
  Interventions: Biological: COVID-19 vaccine
- Rabies vaccine group (Experimental): A total of 120 participants received three doses of rabies vaccine on Day 0, Day 7 and Day 28.
  Blood sampling was performed on Day 0 and Day 42.
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: coadministration — the coadministration of an inactivated COVID-19 vaccine (BBIBP-CorV) and rabies vaccine
  Arms: Co-Ad group
Biological: COVID-19 vaccine — received one dose of inactivated COVID-19 vaccine (BBIBP-CorV)
  Arms: COVID-19 vaccine group
Biological: rabies vaccine — received three dose of rabies vaccine
  Arms: Rabies vaccine group

SUMMARY:
Evaluation of immunogenicity and safety of inactivated COVID-19 vaccine (BBIBP-Cov) coadministered with rabies vaccine.

DETAILED DESCRIPTION:
The participants aged ≥18 who had received two doses of inactivated COVID-19 vaccine were recruited and randomly assigned to one of three study groups: Co-Ad group, COVID-19 vaccine group and Rabies vaccine group.

The participants in Co-Ad group and COVID-19 vaccine group received a booster dose of inactivated COVID-19 vaccine.The participants in Co-Ad group and Rabies vaccine group received three doses of rabies vaccine for pre-exposure immunization. The participants in Co-Ad group received the first dose of rabies vaccine (Day 0) and the inactivated COVID-19 vaccine simultaneously.

Any local or systemic adverse events after vaccination will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18.
* Have the ability to understand the study procedures, voluntarily sign informed consent.
* Be able and willing to complete the entire study plan during the study follow-up period.
* Participants have not received any rabies vaccine.
* Participants have received 2 doses of inactivated COVID-19 vaccine for 6-12 months.
* The time interval between the last vaccination is ≥14 days.
* Body temperature < 37.3 °C confirmed by clinical examination before enrollment .

Exclusion Criteria for the first dose:

* Participants who have received the third dose of COVID-19 vaccine.
* Participants who have previously been infected with COVID-19 or who have tested positive for SARS-CoV-2.
* Having a history or family history of convulsions, epilepsy, encephalopathy and psychosis.
* Being allergic to any component of vaccines and a history of severe allergic reactions to any vaccine.
* Participants are suffering from immunodeficiency, receiving immunosuppressant therapy (oral steroid hormones) during treatment for malignancy, or having low immunity due to HIV within 14 days before enrollment, or having congenital immune disorders in close family members.
* Injection of non-specific immunoglobulin within 1 month before enrollment.
* Participants are suffering from acute febrile diseases and infectious diseases, or have used anti-inflammatory/antiviral/antipyretic/antiallergic drugs within 3 days before enrollment.
* A history of clearly diagnosed thrombocytopenia or other clotting disorders that may contraindicate subcutaneous injection.
* Participants with severe chronic diseases or acute episodes of chronic diseases, hypertension or diabetes that cannot be controlled by drugs.
* Participants with infectious, suppurative and allergic skin diseases.
* Pregnant and lactating women.
* Other Participants whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Exclusion criteria for the second or third dose:

* Participants who had vaccine-related serious adverse reactions after vaccination.
* Systemic adverse reactions/anaphylaxis with severity ≥3 after vaccination as determined by the investigator.
* Participants experienced new conditions that met the "exclusion criteria for the first dose ".
* Other reasons for exclusion considered by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate against SARS-CoV-2 | 28 days after vaccination (Day 28)
  The rate of seroconversion against SARS-CoV-2
Seroconversion rate against rabies virus | 14 days after the 3th dose (Day 42)
  The rate of seroconversion against rabies virus
Neutralizing antibody GMT against SARS-CoV-2 | 28 days after vaccination (Day 28)
  Neutralizing antibody GMT against SARS-CoV-2 after vaccination
Neutralizing antibody GMC against rabies virus | 14 days after the 3th dose (Day 42)
  Neutralizing antibody GMC against rabies virus after 3th dose
Neutralizing antibody GMI against SARS-CoV-2 | 28 days after vaccination (Day 28)
  Neutralizing antibody GMI against SARS-CoV-2 after vaccination
Neutralizing antibody GMI against rabies virus | 14 days after the 3th dose (Day 42)
  Neutralizing antibody GMI against rabies virus after 3th dose

SECONDARY OUTCOMES:
Adverse events rate | 0-7 days or 0-28 days following vaccinations
  Analyse the incidence of adverse events following vaccination, both solicited and unsolicited
Serious adverse event rate | 0-6 months
  Report and analyse serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ruizhi Zhang, Principal Investigator — Guizhou Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Guizhou Provincial Center for Disease Control and Prevention, Guiyang
  - Shanxi Provincial Center for Disease Control and Prevention, Taiyuan

IPD SHARING:
Plan to Share IPD: No